CLINICAL TRIAL: NCT01488747
Title: Bioavailability of Fish Oils: Emulsified vs. Capsular Triglyceride
Brief Title: Bioavailability of Fish Oils: Emulsified Versus Capsular Triglyceride
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GFHNRC023
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Healthy Adults
Keywords: Omega-3 fatty acids; Phospholipid fatty acids; chymlomicron fatty acids; Bioavailability fo fish oil supplements in healthy adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Coromega Omega-3 Squeeze (Experimental): 5.03 g
  Interventions: Dietary Supplement: Coromega Omega-3 Squeeze
- Coromega Nectar (Experimental): 12.22 g
  Interventions: Dietary Supplement: Coromega Nectar
- Barleans Swirl (Experimental): 17.45 g
  Interventions: Dietary Supplement: Barleans Swirl
- Nordic Omega-3 Softgel (Active Comparator): 4 softgels
  Interventions: Dietary Supplement: Nordic Omega-3 Softgel

INTERVENTIONS:
Dietary Supplement: Coromega Omega-3 Squeeze — 660 mg EPA, 434 mg DHA
  Arms: Coromega Omega-3 Squeeze
Dietary Supplement: Coromega Nectar — 660 mg EPA, 436 mg DHA
  Arms: Coromega Nectar
Dietary Supplement: Barleans Swirl — 660 mg EPA, 660 mg DHA
  Arms: Barleans Swirl
Dietary Supplement: Nordic Omega-3 Softgel — 660 mg EPA, 440 mg DHA
  Arms: Nordic Omega-3 Softgel

SUMMARY:
The primary objective of this investigation is to determine the relative percentage and rate of incorporation of eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA) and total omega-3 (n-3) fatty acids after ingestion of 4 emulsified flavored triglyceride fish oil supplements versus an encapsulated triglyceride in defined plasma lipid pools.

The primary endpoints to be evaluated include the fatty acid composition of plasma lipids before and after consumption of a single dose of emulsified triglyceride based fish oil and triglyceride of similar n-3 compositions in capsule form. The investigators will measure changes in plasma phospholipid, and chylomicron fatty acids.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults ages 18 to 60.
2. Body mass index between 22 and 32 kg/m2.
3. Medical history (interview) demonstrating good health.
4. Nonsmoker.
5. Consumption of a typical American diet with no unusual dietary habits.
6. Willingness to comply with the study protocol.
7. Low reported n-3 intake (<100 mg/d) on the Omega-3 Checklist

Exclusion Criteria:

1. Any active, uncontrolled medical problem.
2. Consumption of essential fatty acid supplements within the past 6 months.
3. Use of lipid lowering drugs.
4. Fish consumption greater than 1 fish meal per week

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve for phospholipid fatty acids | 48 hours
  Evaluation of the bioavailability of fatty acids from fish oil supplements

SECONDARY OUTCOMES:
Area under the curve for chylomicron fatty acids | 48 hours
  Evaluation of the bioavailability of fatty acids from fish oil supplements

CONTACTS AND LOCATIONS:
Overall Officials: Susan Raatz, PhD, RD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raatz SK, Redmon JB, Wimmergren N, Donadio JV, Bibus DM. Enhanced absorption of n-3 fatty acids from emulsified compared with encapsulated fish oil. J Am Diet Assoc. 2009 Jun;109(6):1076-81. doi: 10.1016/j.jada.2009.03.006. PMID 19465191
- See also: USDA Grand Forks Human Nutrition Research Center — http://www.ars.usda.gov/main/site_main.htm?modecode=54-50-00-00